CLINICAL TRIAL: NCT02614742
Title: SFX-01 After Subarachnoid Haemorrhage
Acronym: SAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evgen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVG001SAH; 2014-003284-38 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-25 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2019-07

CONDITIONS: Subarachnoid Hemorrhage, Spontaneous
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Cyclodextrins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFX-01 (Active Comparator): 300mg bid for up to 28 days.
  Interventions: Drug: SFX-01
- Placebo (Placebo Comparator): 300mg placebo bid for up to 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SFX-01 — An intervention releasing sulforaphane.
  Other Names: Sulforadex
  Arms: SFX-01
Drug: Placebo — Placebo otherwise identical to Active product
  Other Names: Cyclodextrin
  Arms: Placebo

SUMMARY:
This is a Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of SFX-01 in Subarachnoid Haemorrhage, with exploratory evaluations of efficacy.

DETAILED DESCRIPTION:
The study is a randomised, double-blind, parallel-group design comparing SFX-01 (300 mg) taken orally as capsules or as a suspension via a nasogastric tube (NG) twice-daily for up to 28 days versus placebo in 90 patients who have had SAH and present within 48 hours of ictus.

Subjects will receive SFX-01/Placebo in order to review potential outcomes investigating the long-term complications of SAH such as Delayed Cerebral Ischaemia, as reflected by Trans-Cranial Doppler (TCD) readings. The objective is to demonstrate safety and search for signals of efficacy in patients that have had SAH.

A sub-study will be conducted in up to 12 patients where an External Ventricular Drain (EVD) fitted; serial CSF samples will be taken pre- & post-dose on two occasions to determine pharmacokinetics of Sulforaphane in CSF in comparison with plasma pharmacokinetics. Sub-study patients will undergo all other procedures (with the exception of lumbar puncture).

Treatment duration is up to 28 days; follow up duration is 28 days, three and six months. The planned trial period is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radiological evidence of spontaneous SAH
2. Fisher grade 3 or 4 on CT
3. Definitive treatment of aneurysm has not been ruled out
4. Previously living independently
5. In the opinion of the investigator, the delay from ictus to randomisation and initiation of trial medication will not exceed 48 hours
6. Aged 18 to 80 years
7. In the opinion of the investigator it will be possible to obtain Informed Consent from the Patient, Personal Legal Representative or Professional Legal representative within 24 hours of first dose

Exclusion Criteria:

1. Traumatic SAH
2. Fisher grade 1 or 2
3. SAH diagnosed on lumbar puncture with no evidence of blood on CT
4. Decision not to treat aneurysm has been made
5. Plan to withdraw treatment
6. Significant kidney disease as defined as plasma creatinine ≥2.5mg/dL (221 µmol/l)
7. Liver disease as defined as total bilirubin ≥2-fold the upper limit of normal; (ULN) as measured by the local laboratory
8. Females who are pregnant or lactating.
9. Participants enrolled in another interventional research trial in the last 30 days
10. Patients for whom it is known, at the time of screening, that clinical follow-up will not be feasible Patients unwilling to use two forms of contraception (one of which being a barrier method) 30 days for men and 90 days for women after last IMP dose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Toxicity Criteria | up to 28 days
  To evaluate the safety of up to 28 days of SFX-01 dosed at up to 96 mg Sulforaphane (SFN) per day
Maximum CSF Concentration [Cmax], | up to 28 days
  To detect the presence of SFN in Cerebrospinal Fluid (CSF)
Number of participants with treatment related reduction in middle cerebral artery (MCA) peak flow velocity following Subarachnoid Haemorrhage (SAH) measured by trans cranial doppler ultrasound | up to 28 days
  To determine if a minimum of 7 days treatment with SFX-01 reduces Middle Cerebral Artery (MCA) peak flow velocity following Subarachnoid Haemorrhage (SAH).

SECONDARY OUTCOMES:
modified Rankin Scale | up to 180 days post ictus
  To determine if a minimum of 7 days treatment with SFX-01 improves clinical outcome following SAH as measured using the modified Rankin Scale assessed at 7 , 28, 90 and 180 days post ictus.
Plasma PK | up to 28 days
  To determine plasma SFN levels (and its metabolites) with treatment with SFX-01 (300mg bid).
CSF drug levels | up to 14 days
  To determine CSF drug levels following treatment with SFX-01 (300mg bid).
Serum Haptoglobin levels | Up to 28 days
  To determine if up to 28 days treatment with SFX-01 increases serum haptoglobin (HP) levels following SAH
Delayed Cerebral Ischaemia | Up to 28 days
  To determine if up to 28 days treatment with SFX-01 can reduce the incidence of Delayed Cerebral Ischaemia (DCI) following SAH.

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Bulters, MBChB, BSc, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Southampton General Hospital, Southampton, Hampshire
  - Western General Hospital, Edinburgh
  - The Royal London Hospital, London

REFERENCES:
- [Derived] Zolnourian A, Garland P, Holton P, Arora M, Rhodes J, Uff C, Birch T, Howat D, Franklin S, Galea I, Bulters D. A Randomised Controlled Trial of SFX-01 After Subarachnoid Haemorrhage - The SAS Study. Transl Stroke Res. 2025 Aug;16(4):1031-1043. doi: 10.1007/s12975-024-01278-1. Epub 2024 Jul 19. PMID 39028412
- [Derived] Zolnourian AH, Franklin S, Galea I, Bulters DO. Study protocol for SFX-01 after subarachnoid haemorrhage (SAS): a multicentre randomised double-blinded, placebo controlled trial. BMJ Open. 2020 Mar 25;10(3):e028514. doi: 10.1136/bmjopen-2018-028514. PMID 32217557